CLINICAL TRIAL: NCT04384562
Title: Studying the Role of Brain Molecules for Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020-00044-BEH
Record Dates: First submitted 2020-04-10; First posted 2020-05-12 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Decision Making; Healthy
MeSH Terms: interventions — Methylphenidate; Reboxetine; Nicotine Chewing Gum

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled, between-participant study. In this experiment. Participants will receive a preferential dopamine reuptake inhibitor, a selective noradrenaline reuptake inhibitor, a natural nicotinic acetylcholine receptor agonist, or placebo under double-blind conditions.
Who Masked: Participant, Investigator
Masking Description: All participants will receive the same instructions, and neither they nor the experimenters are informed which drug is used. Participants must take the drug in front of the investigator, to ensure correct intake and compliance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dopamine reuptake inhibitor (Experimental): Participants in the dopamine reuptake inhibitor group will be asked to take one pill containing 20 mg methylphenidate 1.5 hours before the experimental session. One hour later (30 minutes before testing begins), participants will be asked to chew a placebo gum.
  Interventions: Drug: Methylphenidate; Drug: Placebo gum
- Noradrenaline reuptake inhibitor (Experimental): Participants in the noradrenaline reuptake inhibitor group will be asked to take one pill containing 4 mg reboxetine 1.5 hours before the experimental session. One hour later (30 minutes before testing begins), participants will be asked to chew a placebo gum.
  Interventions: Drug: Reboxetine; Drug: Placebo gum
- Cholinergic receptor agonist (Experimental): Participants in the cholinergic receptor agonist group will be asked to take a placebo pill 1.5 hours before the experimental session. One hour later (30 minutes before testing begins), participants will be asked to chew a gum with 2 mg of nicotine.
  Interventions: Drug: Nicotine gum; Drug: Placebo pill
- Placebo (Placebo Comparator): Participants in the placebo group will be asked to take a placebo pill 1.5 hours before the experimental session. One hour later (30 minutes before testing begins), participants will be asked to chew a placebo gum.
  Interventions: Drug: Placebo pill; Drug: Placebo gum

INTERVENTIONS:
Drug: Methylphenidate — A 20 mg methylphenidate (Ritalin®) is administered only once for the dopamine reuptake inhibitor group.
  Other Names: Ritalin®
  Arms: Dopamine reuptake inhibitor
Drug: Reboxetine — A 4 mg reboxetine (Edronax®) is administered only once for the noradrenaline reuptake inhibitor group.
  Other Names: Edronax®
  Arms: Noradrenaline reuptake inhibitor
Drug: Nicotine gum — A 2 mg nicotine (Nicorette®) gum is administered only once for the cholinergic receptor agonist group.
  Other Names: Nicorette®
  Arms: Cholinergic receptor agonist
Drug: Placebo pill — A placebo pill is administered only once.
  Arms: Cholinergic receptor agonist; Placebo
Drug: Placebo gum — A placebo gum is administered only once.
  Arms: Dopamine reuptake inhibitor; Noradrenaline reuptake inhibitor; Placebo

SUMMARY:
The aim of the present project is to elucidate the neuropharmacological mechanisms underlying value (choice preference) and attention (choice randomness) processing in humans. More specifically, the investigators test whether dopaminergic, noradrenergic and cholinergic interventions affect neural and behavioral processing of valuation and attention during decision-making. The investigators do this by up-regulating dopaminergic, noradrenergic or cholinergic neurotransmission pharmacologically through administration of methylphenidate, reboxetine, or nicotine. We test the hypothesis that methylphenidate, reboxetine, or nicotine reduce choice randomness and that this effect is underpinned by an effect on attention and/or value processing.

DETAILED DESCRIPTION:
To simultaneously assess and dissociate choice preference and randomness in stable environments, the investigators plan to use two tasks: (1) a variant of the RISKGARP task, a well-established risky decision-making task and (2) a modified Becker-DeGroot-Marshak task that measures choice preference and the width of preference representations with the range of willingness to pay procedure (range-WTP). Note that wider representations should result in more choice randomness. The investigators will assess choice randomness also by repeating the same decision questions several times within each task and by relating the preferences measured by the RISKGARP task to those measured by the range-BDM task by using the same options in both tasks. To assess the impact of changing environments and learning on choice preference and randomness, participants will perform two established exploration/exploitation tasks. One (3) is a foraging task that has been combined with different pharmacological manipulations and the other (4) is a variant of the four-armed bandit task, which allows distinguishing value- or information-based exploration from random choice. Blood and saliva samples may be taken. Blood samples may be used to determine levels of the administrated substances and to assess genetic variation. Saliva samples may be used to determine cortisol and testosterone levels.

ELIGIBILITY:
Inclusion Criteria:

* Physically and psychiatrically healthy (as defined by exclusion criteria) men and women aged 18-35 years
* Ability and willingness to participate in the study
* Willingness to not eat or drink any food/beverage containing caffeine or alcohol 12 hours prior to the administration of study medication (asked in screening session)
* Willingness to not eat or drink grapefruit or grapefruit related citrus fruits (e.g., Seville oranges, pomelos) from 7 days prior to the administration of study medication (asked in screening session)
* Good command of English language (be able to understand the task instructions and in the unlikely case of adverse effects inform the examiner)
* Signed informed consent

Exclusion Criteria:

* Serious past brain disease or injury
* Frequent headaches (of any sort, > 1/week) or migraine (irrespective of frequency)
* History of epileptic seizures
* Any neurological disorder
* Surgery to head or heart (MRI safety, potential metal pieces)
* Pacemaker, hearing aid or neurostimulator (MRI safety, metal pieces)
* Known cardiac or cardiovascular disease or anomaly
* Family history of sudden death due to cardiac arrhythmia
* High or low blood pressure, history of heart attack, infrequent heartbeat
* Respiratory problems (including difficulty with breathing through the nose)
* Glaucoma (present or past)
* Insufficiency of kidney or liver, acute liver disease
* Any psychiatric disorder (especially depression, mania, schizophrenia, addiction panic and suicidality)
* Severe vocal or motor tics (methylphenidate, data quality)
* Severe psychosomatic disorder (somatic complaints without clear medical cause, has a mental component)
* Potential metal parts in body (MRI safety; metal splinters, gun wounds, shrapnel or surgical clips)
* Pregnancy, nursing, or currently planned pregnancy
* Allergy to drugs, particularly methylphenidate, reboxetine or nicotine
* Severe intolerance to lactose including strong diarrhea after only a few mg (weak lactose intolerance is no exclusion criterion as medication only contains a very small dose (around 4 mg) of lactose)
* Oversensitivity to hot pepper sauce (e.g., tabasco)
* Currently taking any medication or recently participated in other clinical trials that might interfere with Methylphenidate and Reboxetine, especially MAO-Inhibitors (e.g. Aurorix (Moclobemid) and Azilect (Rasagilin), antipsychotics, antibiotics, and medication for heart diseases
* Currently taking any further medication (besides birth control) or natural products (infrequent intake of natural products and/or food supplements need to be mentioned to the examiner)
* Drug abuse (exclude people with a positive test)
* Serious acute or chronic disease that could interfere with participation in the experiments
* Inability to lie still in the scanner (e.g. due to itching, sneezing, coughing, claustrophobia)
* Inability to understand the instructions
* Participants with BMI < 18
* Clinically relevant score in STAI T (anxiety), measured during screening on a separate day
* ECG demonstrating QTcF >450 msec or a QRS interval >120 msec at screening. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTcF/QRS values should be used to determine participant eligibility, measured during screening on a separate day
* Participants who eat or drink grapefruit or grapefruit related citrus fruits (e.g., Seville oranges, pomelos) or drinks from 7 days prior to the administration of study medication.
* Participants who eat or drink any food/beverage containing caffeine or alcohol 12 hours before the study
* Current smokers/tobacco consumers (exclude people whose cotinine level is higher than 50ng/ml with a urine test)
* Phenylketonuria
* Dental or jaw condition prohibiting gum chewing
* Pheochromocytoma
* Thyroid disorders
* Diabetes
* Type of angina where chest pain occurs at rest
* Unpredictable severe constricting chest pain
* Prickling or tingling of fingers and toes
* Buerger's Disease
* Throat irritation
* Peptic ulcers
* Esophagitis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Choice data | All participants perform decision-making tasks after drug/placebo administration in the main experimental session lasting about 1 hour.
  Choice data made by participants are measured from the experimental tasks. More specifically, the investigators calculate choice preferences, such as the percentage of trials in which participants chose options with probabilistic outcomes in the RISKGARP task and the bids they made in the Range-WTP task, the percentage of exploitative/explorative choices in the four-armed bandit task, and the leaving time in the foraging task. Moreover, the investigators determine choice sub-optimality, such as the number of choices violating transitivity in the RISKGARP task, the inconsistency of bids in repeated trials in the Range-WTP task, the percentage of selecting the worst option in the four-armed bandit task, and the difference between optimal leaving time and actual leaving time in the foraging task.
Response time data | All participants perform decision-making tasks after drug/placebo administration in the main experimental session lasting about 1 hour.
  Response times are measured from experimental tasks. The investigators calculate how long participants take to make decisions in each trial.

SECONDARY OUTCOMES:
The size of pupil dilation | Pupil size is measured in the main experimental session before drug/placebo administration and through study completion lasting about 1 hour.
  Pupil size is measured using eye-tracker while participants perform the experimental tasks. Baseline pupil size is also measured before the drug/placebo administration.

OTHER OUTCOMES:
Computational parameters estimated from experimental data | All participants perform decision-making tasks after drug/placebo administration in the main experimental session lasting about 1 hour.
  Computational parameters are estimated from the data of participants during the decision-making tasks. Specifically, mathematical models will be applied to above-mentioned choice data and/or response time data. The estimated parameters reflect choice preference and stochasticity and are complementary to the descriptive measurements mentioned above. For example, utility functions will be estimated and the choice preferences are described by the concavititvity of utility functions.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Tobler, PhD, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Doren N, Chung HK, Grueschow M, Quednow BB, Hayward-Konnecke H, Jetter A, Tobler PN. Acetylcholine and noradrenaline enhance foraging optimality in humans. Proc Natl Acad Sci U S A. 2023 Sep 5;120(36):e2305596120. doi: 10.1073/pnas.2305596120. Epub 2023 Aug 28. PMID 37639601